CLINICAL TRIAL: NCT06097715
Title: Clinical, Endoscopic and Radiological Assessment of Portal Hypertension in Children With Chronic Liver Diseases
Brief Title: Clinical,Endoscopic and Radiological Assessment of Portal Hypertension in Children With Chronic Liver Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Abuelfadl, specialist of pediatrics at sohag teaching hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-10-02MD
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient group (Active Comparator): patients which previosly diagnosed with chronic liver diseases or presented with manifestations of chronic liver diseases
  Interventions: Diagnostic Test: upper gastrointestinal endoscopy; Diagnostic Test: 1- Complete blood count 2- Coagulation profile
- control group (Active Comparator): children in the same age and sex of the patient group and presented to Sohag Universty Hospital due to any complaint rather than hepatic and gastrointestinal disease.
  Interventions: Diagnostic Test: 1- Complete blood count 2- Coagulation profile

INTERVENTIONS:
Diagnostic Test: upper gastrointestinal endoscopy — Upper gastrointestinal endoscopy to asses present of esophageal varices and will be done to all patient group
  Arms: patient group
Diagnostic Test: 1- Complete blood count 2- Coagulation profile — cmplete blood count to detect thrombocytopenia, liver function test to detect if they are elevated,and any impaired coagulation profile

SUMMARY:
Portal hypertension is a significant cause of morbidity and mortality in children with chronic liver disease and portal vein obstruction. It results in severe complications such as ascites, hepatic encephalopathy and gastrointestinal variceal bleeding. (Sutton et. al., 2018).

Esophageal varices is an important manifestation of portal hypertension that develops over time in children with chronic liver disease. The risk of esophageal varices hemorrhage increases depending on the underlying disease as well as the duration of the disease and the mortality rate as high as 5% - 20 % during patient follow up. Invasive procedures such as gastroscopy are performed repeatedly to detect the presence and progression of esophageal varices. Many non-invasive methods have been investigated to their efficacy in determining the presence of esophageal varices and the risk of complications in the presence of portal hypertension. (Taşkın et.al., 2023).

Early diagnosis of portal hypertension is often difficult as it can be asymptomatic. During this stage, the patient may feel nothing except for mild fatigue or abdominal discomfort and therefore, patients mostly go undiagnosed (Hartl et.al., 2021). (Selicean et.al., 2021). However, it is worth noting that some of the results from medical investigation may be abnormal during this stage. These include abnormal liver function, abnormal routine blood examination (thrombocytopenia), and changes in the stiffness of the liver which can be found during ultrasound despite the patient being asymptomatic. ( Mohanty et al., 2021).

Though the gold standard to diagnose portal hypertension is hepatic venous pressure gradient (HVPG) and a value more than 10 mmHg defines clinically significant portal hypertension (CSPH) ( Man Zhang et.al., 2022). Since HVPG measurement is scarcely available and invasive, several non-invasive tests are used as surrogate markers of CSPH. Amongst them, elastography techniques measuring liver stiffness (LS) and spleen stiffness (SS) are the extensively studied ones which can be done by elastography machines that can be attached to conventional ultrasound (USG) machines . Amongst them, 2D-shear wave elastography (2D-SWE) is the most recent one, and it assesses stiffness and related parameters by tracking shear waves propagated through a media. (Sattanathan et.al., 2023).

ELIGIBILITY:
Inclusion Criteria:

- 1- Age: < 18 years 2- Manifestations of hepatic disease like jaundice, hepatic encephalopathy, organomegally.

3- Children previously diagnosed with chronic liver disease

Exclusion Criteria:

* 1- Age: > 18 years. 2- Non compliant child during technique of elastography. 3- Patient with ascites. 4- Patient with portosystemic shunt surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with early detection of portal hypertension in patient with chronic liver diseases | 1 year
  we aim to early of portal hypertension in patient with chronic liver diseases before occurance of complications as esophageal bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sutton H, Dhawan A, Grammatikopoulos T. Non-invasive Markers of Portal Hypertension: Appraisal of Adult Experience and Potential Utilisation in Children. J Pediatr Gastroenterol Nutr. 2018 Apr;66(4):559-569. doi: 10.1097/MPG.0000000000001882. PMID 29287004
- [Background] Zhang M, Jin H, Cao J, Ren R, Jia M, Yang Y, Li X, Chen M, Li S, Huang L, Ling W. Application of Ultrasound Elastography in Assessing Portal Hypertension. Diagnostics (Basel). 2022 Sep 29;12(10):2373. doi: 10.3390/diagnostics12102373. PMID 36292062
- [Background] Hartl L, Jachs M, Desbalmes C, Schaufler D, Simbrunner B, Paternostro R, Schwabl P, Bauer DJM, Semmler G, Scheiner B, Bucsics T, Eigenbauer E, Marculescu R, Szekeres T, Peck-Radosavljevic M, Kastl S, Trauner M, Mandorfer M, Reiberger T. The differential activation of cardiovascular hormones across distinct stages of portal hypertension predicts clinical outcomes. Hepatol Int. 2021 Oct;15(5):1160-1173. doi: 10.1007/s12072-021-10203-9. Epub 2021 May 21. PMID 34021479
- [Background] Selicean S, Wang C, Guixe-Muntet S, Stefanescu H, Kawada N, Gracia-Sancho J. Regression of portal hypertension: underlying mechanisms and therapeutic strategies. Hepatol Int. 2021 Feb;15(1):36-50. doi: 10.1007/s12072-021-10135-4. Epub 2021 Feb 5. PMID 33544313